CLINICAL TRIAL: NCT00677430
Title: Multimodality Anthropometric Analysis for Quantitative Assessment of Outcomes in Breast Reconstructive Surgery
Brief Title: Quantitative Analysis of Outcomes in Breast Reconstruction
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2004-0899; RSGPB-09-157-01-CPPB (Other Grant/Funding Number: American Cancer Society)
Record Dates: First submitted 2008-05-09; First posted 2008-05-14 (Estimated); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Breast Reconstruction; Digital Imaging; Questionnaire; Survey
MeSH Terms: conditions — Breast Neoplasms | interventions — Surveys and Questionnaires; Quantitative Phase Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Questionnaire + Digital Imaging: A brief questionnaire packet will be completed. Photographs of the breast(s) will be taken with two different types of digital cameras (2D and 3D). The photos will be used to develop automated methods for evaluating the appearance and shape of the breasts.
  Interventions: Behavioral: Questionnaire; Procedure: Digital Imaging

INTERVENTIONS:
Behavioral: Questionnaire — A brief questionnaire packet will be completed.
  Other Names: Survey
Procedure: Digital Imaging — Photographs of the breast(s) will be taken with two different types of digital cameras (2D and 3D). The photos will be used to develop automated methods for evaluating the appearance and shape of the breasts.

SUMMARY:
The first objective of this study is to assess the accuracy of digital image-processing techniques to provide measurements of human breast physical dimensions. The ultimate usefulness of these techniques is to develop quantitative outcome measures of the visual appearance of breast after local treatments for breast cancer. These measures will be used to improve clinical outcomes from multimodality therapy that includes surgery and radiotherapy and form the basis for the future development of patient decision making aids. The second objective is to evaluate the relationship between patient reported body image outcomes and measurement of human breast physical dimensions for patients with breast cancer.

DETAILED DESCRIPTION:
If you agree to take part in this study, you will be asked to fill out a brief questionnaire packet. This packet contains questions about how you feel about your appearance and your overall well-being. You will be asked to have photographs of your breast(s) taken with two different types of digital cameras (2D and 3D). These are the same type of photographs routinely taken for all patients having breast reconstructive surgery. The photographs and measurements will be taken during your routine clinic visit. You will not be identifiable in the photographs.

The photographs will be used to develop automated methods for evaluating the appearance and shape of the breasts.

You may be asked to complete additional follow-up visits for this study. These visits would take place at a regularly-scheduled clinic visit that takes place just before a surgical procedure is planned. At these visits you would be asked to fill out another questionnaire packet and to allow the research the research staff to repeat the photographs. The number of follow-up visits needed would depend on your individual treatment plan. A final study visit would take place once you feel you are finished with your breast reconstructive process. At this point, your participation in the study would be completed. Breast reconstruction is different for each patient. The length of time of the reconstructive process depends on the procedure(s) that you and your surgeon have agreed upon. These options will be discussed at your regularly scheduled clinic appointments.

This is an investigational study. A total of up to 300 patients will take part in this study. All will be enrolled at UTMDACC.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. Age greater than 21 years old.
3. Candidate who has had or is planning to have breast reconstructive surgery and has at least one breast mound.
4. Willing to participate in the study and able to complete informed consent.
5. Proficient at reading and speaking English.

Exclusion Criteria:

1. Women who have undergone previous bilateral mastectomy without reconstruction.
2. Women who are unable to stand unassisted for 2 minutes.
3. Diagnosis of serious mental illness (e.g. schizophrenia) or cognitive impairment.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants with breast cancer that have had or are about to have breast reconstructive surgery.
Sampling Method: Non-Probability Sample
Enrollment: 224 (Actual)
Dates: Start 2008-05 (Actual); Primary Completion 2021-04-09 (Actual); Study Completion 2021-04-09 (Actual)

PRIMARY OUTCOMES:
Evaluate accuracy of digital image-processing techniques used to provide the physical dimensions of human breasts. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Gregory P. Reece, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org